CLINICAL TRIAL: NCT01916265
Title: A Randomised, Single Center, Three-period Trial to Compare the Relative Pharmacodynamic Properties of Different Glucagon Dosages at Four Different Blood Glucose Concentrations
Brief Title: Trial to Compare the Relative Pharmacodynamic Properties of Different Glucagon Dosages
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PCDiab01
Record Dates: First submitted 2013-07-25; First posted 2013-08-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Glucagon

ARMS (3):
- Glucagon level: 0,11 and 1 mg (Experimental): Glucagon level: 0,11 and 1 mg
  Interventions: Drug: Glucagon
- Glucagon level: 0,22 and 0,66 mg (Experimental): Glucagon level: 0,22 and 0,66 mg
  Interventions: Drug: Glucagon
- Glucagon level: 0,44 and 0,33 mg (Experimental): Glucagon level: 0,44 and 0,33 mg
  Interventions: Drug: Glucagon

INTERVENTIONS:
Drug: Glucagon

SUMMARY:
The ultimate goal of the PCDIAB project is to develop a bi-hormonal pump (insulin and glucagon) substituting for the pancreas and facilitating tight euglycemic control in patients with T1DM.

DETAILED DESCRIPTION:
The study is planned as open, randomised 3-period cross-over in patients with T1DM. The study will include a total of 6 completing patients. The study is not blinded due to the exploratory nature.

At each of the 3 periods, different blood glucose level will be established in 4 steps (8, 6, 4, and 2.8 mmol/L), and a prefixed glucagon dose will be given per glucose level. The sequence of glucagon dose strength for the three dosing days will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with diabetes mellitus type 1 , as defined by the American Diabetes Association1.
* Age ≥ 18 and ≤ 65 years.

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products.
* Receipt of any investigational medicinal product within 3 months or 5 half-lives of that IMP before randomisation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
AUCGlucose of different glucagon dosages given s.c. | 90 min after dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany